CLINICAL TRIAL: NCT07402031
Title: Research of Predictive Factors of Weight Loss After Bariatric Surgery in Patients Suffering From Obesity
Brief Title: Predicting Weight Loss After Bariatric Surgery in Patients With Obesity
Status: Not yet recruiting | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: TCAPrediBaria
Record Dates: First submitted 2026-01-13; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Bariatric Surgery
MeSH Terms: interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Bariatric surgery — Longitudinal follow-up of participants whose application for bariatric surgery was accepted. It will combine anthropometric, clinical, neuropsychological and biological measurements taken at various timepoints. Participants will be asked to complete a set of online questionnaires and data will be recorded anonymously. Biological samples will be collected at various time points.

SUMMARY:
As with other nutritional strategies, the clinical response to bariatric surgery can be highly variable, with weight regain being a frequent occurrence. Among multiples factors, co-occurrence of eating disorders such as binge eating disorder has been implicated in insufficient clinical response. Improving our ability to predict how patients will respond to surgery is necessary in order to tailor the care pathways we offer. The mechanisms involved in disturbances of eating behaviour before and after surgery remain largely unknown. This study aims to identify the predictive factors of weight loss after bariatric surgery, as well as the cognitive and biological mechanisms that mediate this effect.

ELIGIBILITY:
Inclusion criteria:

* Age between 18 and 65 years
* Obesity, with bariatric surgery indicated after a multidisciplinary evaluation.
* Good physical and mental health, enabling informed consent.
* French speaker

Exclusion criteria:

* Legal protection
* Pregnancy or breastfeeding
* History of bariatric surgery (except gastric banding, provided it was removed more than five years ago).
* Acute or progressive chronic disease
* Alcohol consumption of more than 20 g/day
* Inflammatory bowel disease;
* Digestive autonomic diabetic neuropathy.
* Consumption of dietary supplements (stanols, probiotics, prebiotics or omega-3).
* Following a vegan or gluten-free diet or being lactose intolerant.
* Fibre consumption >30 g/day
* Recent change in antidiabetic medication within the past 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants candidates for bariatric surgery once its indication has been validated by a multidisciplinary committee, following medical, nutritional and psychological evaluations.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2032-06 (Estimated); Study Completion 2036-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between weight loss after surgery and clinical, neuropsychological and biological parameters. | Throughout the entire study, aproximately during 5 years
  The percentage of excessive weight loss after bariatric surgery will be correlated with
  * Clinical parameters (Binge Eating Scale and modified Yale Food Addiction Scale 2.0)
  * Neuropsychological parameter (Barratt Impulsivness Scale and Trail Making Test)
  * Biological parameters

SECONDARY OUTCOMES:
Binge Eating Disorder. | Throughout the entire study, aproximately during 5 years
  Evaluation of eating disorders using the Binge Eating Scale (BES).
Food Addiction. | Throughout the entire study, aproximately during 5 years
  Evaluation of food addiction will be performed using modified Yale Food Addiction Scale 2.0.
Eating attitudes | Throughout the entire study, aproximately during 5 years
  Eating patterns and habits will be screened using the Eating Attitude Test 26
Cognitive flexibility. | Throughout the entire study, aproximately during 5 years
  Neuropsychological evaluation of cognitive flexibility will be performed with the Trail Making Test
Impulsivity. | Throughout the entire study, aproximately during 5 years
  Impulsivity will be assessed using the Barrat Impulsiveness Scale (BIS)
Self-reported quality of life. | Throughout the entire study, aproximately during 5 years
  Self-reported quality of life will be assessed using the QOLOD (Quality of Life, Obesity and Dietetics)
Obesity. | Throughout the entire study, aproximately during 5 years
  Weight will be measured at each timepoint
Physical activity. | Throughout the entire study, aproximately during 5 years
  Weekly physical activity will be reported with the Godin Leisure Time Exercise Questionnaire (GLTEQ)
Food intake. | Throughout the entire study, aproximately during 5 years
  Eating habits will be recorded with a Food Frequency Questionnaire (FFQ)
Blood samples | Throughout the entire study, aproximately during 5 years
  Blood samples will be collected and processed for metabolomic analyses.
Fecal sample | Throughout the entire study, aproximately during 5 years
  Feces samples will be collected and processed to evaluation gut-microbiota composition

OTHER OUTCOMES:
Sociodemographic data | Once at inclusion
  Number of children and marital status will be recorded
Medical history | Once at inclusion
  Information concerning medical comorbidities will be collected from the patient medical record.
Childhood Trauma. | Once at inclusion
  Assessment of adverse life events and trauma will used the Childhood Trauma Questionnaire - short form.

CONTACTS AND LOCATIONS:
Overall Officials: Amandine Everard, Professor, Study Director — Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No